CLINICAL TRIAL: NCT01188460
Title: A Cognitive-Behaviour Therapy (CBT) Self-Management Approach for Insomnia in Chronic Pain: A Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Ottawa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009902
Record Dates: First submitted 2010-08-19; First posted 2010-08-25 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2017-08

CONDITIONS: Insomnia; Chronic Pain
Keywords: Insomnia; Chronic pain
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Placebo Comparator): Receive one weekly telephone follow-up call per week to monitor sleep progress, complete 7 weeks of sleep diaries only (sleep diary measures Total Sleep Time in hours, Time to Fall Asleep in minutes, Number of Nocturnal Awakenings, Sleep Efficiency as a percentage, and Sleep Quality as units on a scale), complete questionnaires at three study timepoints
  Interventions: Behavioral: Sleep diary
- Experimental Group (Experimental): Receive one weekly telephone call to monitor sleep progress, complete 7 weeks of sleep diaries (sleep diary measures Total Sleep Time in hours, Time to Fall Asleep in minutes, Number of Nocturnal Awakenings, Sleep Efficiency as a percentage, and Sleep Quality as units on a scale), implement one chapter per week of self-help manual for insomnia over 7 weeks at home, complete questionnaires at three study timepoints
  Interventions: Behavioral: Self-help manual for insomnia; Behavioral: Sleep diary

INTERVENTIONS:
Behavioral: Self-help manual for insomnia — Implementation of chapters of self-help manual at home, and completion of sleep diary in terms of time in bed, hours of sleep, time to fall asleep, number of awakenings, and sleep quality
  Other Names: Intervention Group
  Arms: Experimental Group
Behavioral: Sleep diary

SUMMARY:
This study will test the impact of a cognitive-behavioural self-management approach for the management of insomnia among patients with chronic pain. This self-management approach consists of a manual describing cognitive behavioural techniques for the management of insomnia. In terms of primary outcomes, it is anticipated that there would be improvements in sleep-related dimensions such as sleep quality, sleep efficiency, and night-time awakenings in the sample group receiving a copy of the self-help manual intervention to be implemented by participants in their home (intervention group), relative to the group receiving treatment as usual (control group). In terms of secondary outcomes, it is anticipated that the intervention group will show improvements in mood, fatigue, pain severity, and pain-related disability relative to the control group. The tertiary outcome variable of pre-sleep arousal is anticipated to have a moderating or mediating relationship with the sleep variables investigated.

DETAILED DESCRIPTION:
In summary therefore, insomnia and other sleep difficulties have been reported to frequently occur in conjunction with other medical or psychiatric disorders, however insomnia co-occurring with other medical or psychiatric conditions has received less attention relative to primary insomnia with no such concurrent conditions (e.g., Lichstein, 2006; McCrae, & Lichstein, 2001; Taylor, Mallory, Lichstein, Durrence, Riedel, & Bush, 2007). In chronic pain, there have not been many well-controlled studies involving insomnia existing with a concurrent chronically painful condition. Research thus far has found multi-component cognitive-behavioural approaches to be successful in treating primary insomnia, and there have been some studies applying these approaches in the context of insomnia and concurrent medical conditions (Currie, Wilson, Pontefract, & deLaplante, 2000; Morin, 1993). Based on Morin's work (Morin, 1993; Morin, Beaulieu-Bonneau, LeBlanc, & Savard, 2005) involving a cognitive-behaviour therapy (CBT) protocol for patients with sleep problems related to chronic pain, a self-help format of such an intervention has also been developed (Currie & Wilson, 1997). However, this has thus far only been delivered within a group-based treatment programme (Currie, 1998; Currie & Wilson, 1997; Currie, Wilson, Pontefract, & deLaplante, 2000). From this context, and building on a prior study involving a group treatment format (Currie, 1998; Currie, Wilson, Pontefract, & deLaplante, 2000), the usefulness of a manualized self-management approach in manageing insomnia will be investigated, including the impact of this approach with regard to other salient measures of improved functioning (such as pain severity or pain-related disability) for individuals with chronic pain. The proposed study will involve a randomized control trial of this self-help treatment strategy for comorbid insomnia in chronically painful medical conditions among an adult outpatient sample at a hospital rehabilitation centre and pain clinic. This study thus seeks to investigate how successful a cognitive-behaviour therapy (CBT) self-help management approach is for manageing insomnia amongst people with chronic pain. Given the public health implications of the relationship of poor sleep to quality of life (e.g., Morin, Stone, McDonald, & Jones, 1994; Quesnel, Savard, Simard, Ivers, & Morin, 2003), a self-management approach to insomnia in the context of chronic pain may offer an accessible and cost-effective treatment option.

The following hypotheses will be tested:

The first hypothesis predicts that participants in the intervention group will show changes in their scores on psychological measures in terms of greater improvements in sleep-related dimensions, in comparison with controls between the baseline and post-treatment periods.

The second hypothesis predicts that participants in the intervention group will show changes in their scores on psychological measures in terms of lower levels of anxiety, depression, fatigue, pain severity, and pain-related disability, in comparison with controls between the baseline and post-treatment periods. These secondary outcome variables are not directly targeted by the intervention, however it is proposed that if improvements in sleep are experienced, there would be subsequent improvements in the variables of mood, fatigue, pain severity, and pain-related disability among chronic pain patients who experience insomnia.

The third hypothesis predicts that the variable of pre-sleep arousal will have a moderating or mediating influence on the sleep-related variables (which will be the primary outcome variables). The moderating or mediating variable of pre-sleep arousal is proposed to assess dimensions related to sleep that are not tapped into by the primary outcome, sleep-related variables, but that may be of salience in the context of insomnia that is comorbid with chronically painful conditions.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age
* Not in state of crisis
* Able to read and understand English
* Experiences sleep difficulties or insomnia
* Has chronic pain

Exclusion Criteria:

* Under 18 or over 65 years of age
* In a state of crisis
* Does not read or understand English
* Does not experience sleep difficulties or insomnia
* Does not have chronic pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-04; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith E Wilson, PhD, Principal Investigator — The Ottawa Hospital Rehabilitation Centre
Locations (2):
- Canada (2):
  - The Ottawa Hospital, Pain Clinic, Ottawa, Ontario
  - The Ottawa Hospital Rehabilitation Centre, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Receive one weekly telephone follow-up call per week to monitor sleep progress, complete 7 weeks of sleep diaries only, complete questionnaires at three study timepoints
  Sleep diary: Completion of sleep diary in terms of time in bed, hours of sleep, time to fall asleep, number of awakenings, and sleep quality
- Experimental Group: Receive one weekly telephone call to monitor sleep progress, complete 7 weeks of sleep diaries, implement one chapter per week of self-help manual for insomnia over 7 weeks at home, complete questionnaires at three study timepoints
  Self-help manual for insomnia: Implementation of chapters of self-help manual at home, and completion of sleep diary in terms of time in bed, hours of sleep, time to fall asleep, number of awakenings, and sleep quality
Period: Overall Study
Arm/Group | Control Group | Experimental Group
Started | 25 | 23
Completed | 25 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Experimental Group | Total
Number analyzed (Participants) | 25 | 23 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Missing data for age for one participant
  years
    number analyzed (Participants) | 24 | 23 | 47
    (all) | 44.29 (9.55) | 47.96 (10.21) | 46.09 (9.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity Index (ISI)
Description: Measures insomnia symptoms, scores range from 0-28 with higher scores (ranging from 15-28) indicating clinical insomnia and therefore worse outcomes
Time Frame: Timepoint 2 (week 7 of study participation)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 25 | 23
units on a scale | 19.84 (4.14) | 16.04 (5.16)

2. Primary Outcome: Sleep Diary- Total Sleep Time
Description: Measures:
  Total Sleep Time in hours, higher scores indicate better outcomes
Time Frame: Timepoint 2 (week 7 of study participation).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 25 | 23
hours | 5.34 (1.12) | 5.46 (1.02)

3. Primary Outcome: Sleep Diary- Time to Fall Asleep
Description: Measures:
  Time to Fall Asleep in minutes, higher scores indicate worse outcomes
Time Frame: Timepoint 2 (week 7 of study participation).
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 25 | 23
minutes | 0.46 (0.23) | 0.35 (0.15)

4. Primary Outcome: Sleep Diary- Number of Nocturnal Awakenings
Description: Measures:
  Number of Nocturnal Awakenings, higher scores indicate worse outcomes
Time Frame: Timepoint 2 (week 7 of study participation).
Measure: Mean (Standard Deviation); unit: Number of nocturnal awakenings
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 25 | 23
Number of nocturnal awakenings | 3 (1) | 3 (1)

5. Primary Outcome: Sleep Diary- Sleep Efficiency
Description: Measures:
  Sleep Efficiency (percentage)- higher scores indicate better outcomes
Time Frame: Timepoint 2 (week 7 of study participation).
Measure: Mean (Standard Deviation); unit: Percentage of efficiency
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 25 | 23
Percentage of efficiency | 63.06 (8.33) | 67.09 (8.37)

6. Primary Outcome: Sleep Diary- Sleep Quality
Description: Measures:
  Sleep Quality (units on a scale from 0-10), higher scores indicate better outcomes
Time Frame: Timepoint 2 (week 7 of study participation).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 25 | 23
units on a scale | 4 (1) | 4 (1)

7. Secondary Outcome: Pain Severity Rating
Description: Measures pain severity, rated on scale from 0-10, total scores range from 0-40, higher scores indicate worse outcomes
Time Frame: Timepoint 2 (week 7 of study participation).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 25 | 23
units on a scale | 27.96 (5.19) | 25.35 (6.93)

8. Secondary Outcome: Pain Disability Index (PDI)
Description: Measures pain disability impact on various life domains, scores range from 0-70, higher scores indicate worse outcomes
Time Frame: Timepoint 2 (week 7 of study participation).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 25 | 23
units on a scale | 48.12 (11.46) | 46.13 (10.76)

9. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS)
Description: Measures symptoms of depression and anxiety, total scores range from 0-42, higher scores indicate worse outcomes
Time Frame: Timepoint 2 (week 7 of study participation).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 25 | 23
units on a scale | 22.08 (7.43) | 19.43 (5.32)

10. Secondary Outcome: Pre-Sleep Arousal Scale (PSAS)
Description: Measures pre-sleep hyperarousal, total scores range from 16-80, higher scores indicate worse outcomes
Time Frame: Timepoint 2 (week 7 of study participation).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 25 | 23
units on a scale | 44.84 (11.52) | 35.43 (9.14)

11. Secondary Outcome: Fatigue Severity Scale (FSS)
Description: Measures symptoms of fatigue, total scores range from 9-63, higher scores indicate worse outcomes
Time Frame: Timepoint 2 (week 7 of study participation).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 25 | 23
units on a scale | 50.60 (8.74) | 47.30 (10.12)

ADVERSE EVENTS:
Arm/Group | Control Group | Experimental Group
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/23
Other Adverse Events (participants affected / at risk) | 0/25 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes